CLINICAL TRIAL: NCT05423821
Title: Out Patient Anesthesia Experiences in Pediatric Magnetic Resonance Imaging Cases
Brief Title: Non-operating Room Anesthesia Experiences in Pediatric Magnetic Resonance Imaging Cases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yunus Emre (Other)
Responsible Party: Sponsor-Investigator, Yunus Emre, SPECIALIST DOCTOR, Ankara Training and Research Hospital
Organization: Ankara Training and Research Hospital (Other)
Other Study IDs: ytuncdemir-MR
Record Dates: First submitted 2022-06-13; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Magnetic Resonance Imaging Contrast Media Adverse Reaction; Sedation Complication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Anesthesia efficacy in patients undergoing MRI — atropine will be administered when bradycardia develops, oxygen will be given if hypoxia develops

SUMMARY:
In recent years, out patient anesthesia applications have been increasing for diagnostic and interventional procedures for pediatric patients. In this study, we aimed to retrospectively analyze the anesthesia applications performed in pediatric MRI cases in our hospital.

It is a retrospective study

DETAILED DESCRIPTION:
In recent years, applications with sedation and/or general anesthesia for diagnostic purposes in pediatric cases with Magnetic Resonance Imaging (MRI) method have been increasing. Although imaging methods are useful in diagnosis and treatment, they carry minimal risk for patients. As the demands for anesthesia increase during Magnetic Resonance Imaging, questions have arisen about what can be done safely in anesthesia management. The type of anesthesia applied for Magnetic Resonance Imaging is called non-operating room anesthesia.

Cross-sectional imaging techniques such as MRI require pediatric patients to remain calm for up to one hour, and thus these patients need anesthesia. In the induction of anesthesia with agents used in anesthesia outside the operating room, the patient sleeps quickly, the vital functions are stable in its maintenance, the patient recovers quickly after anesthesia, the physical and mental activities return to normal as soon as possible after recovery, and there are no side effects such as nausea, vomiting, dizziness and pain that will delay the discharge. is necessary. Sedation or general anesthesia carries risks and can have unintended consequences if poorly managed.

ELIGIBILITY:
Inclusion Criteria:

* Elective cases under the age of 18 will be included in the study between 01.01.2020 and 01.01.2022.
* Patients to undergo elective magnetic resonance imaging

Exclusion Criteria:

* Magnetic resonance without anesthesia will not be included. Over the age of 18 will be excluded from study

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Cases under the age of 18 who received anesthesia outside the operating room (MRI) in our clinic between 2020-2022 will be screened retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-06-14 (Estimated); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-07-25 (Estimated)

PRIMARY OUTCOMES:
The type of anesthesia we trust most in magnetic resonance | two hour
  genel anesthesia

SECONDARY OUTCOMES:
reducing complications in magnetic resonance | two hour
  mechanical ventilator, endtidal carbon dioxide, non-invasive oxygen saturation

IPD SHARING:
Plan to Share IPD: Undecided